CLINICAL TRIAL: NCT03116633
Title: An Observational Multicenter Study to Evaluate the Performance and Utility of Inivata Liquid Biopsy Analysis Compared With Tissue Biopsy Analysis for Detection of Genomic Alterations in Patients With Lung Cancer
Brief Title: Concordance of Inivata Liquid Biopsy With Standard Tissue Biopsy
Status: Completed | Type: Observational
Sponsor: Inivata (Industry)
Collaborators: Guardian Research Network, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: GRN-ALV
Record Dates: First submitted 2017-04-05; First posted 2017-04-17 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: lung cancer; biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm A: 1st line setting-approx. 150 patients. collect tissue biopsy per standard of care & one blood draw (40ml)
- Arm B: 1st line setting- approx. 100 patients one blood draw (40ml)
- Arm C: Approx. 10 patients tissue collection optional 3 blood draws (40ml) over 5 days

SUMMARY:
This study aims to look at a comparison of liquid biopsy (blood sample) analysis compared with tissue biopsy in patients with advanced lung cancer

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the concordance of Inivata liquid biopsy panel with standard tissue biopsy analysis for detecting genomic alterations in patients with advanced non-squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent
* Male & female patients aged 18 years and over diagnosed with stage IIIb/IV non-squamous NSCLC.
* Patients intended to initiate first-line treatment (Arms A and B)
* Patients who plan to have or have had a recent tumor tissue biopsy taken as part of their standard of care (Arm A)
* Patient must understand and be able, willing and likely to fully comply with all study procedures and restrictions.

Exclusion Criteria:

* Patients who have received any approved or experimental cancer therapy since their most recent NSCLC tissue biopsy
* Any history of metastatic cancer.
* Previous malignancy in the last 2 years (except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix).
* Patient with a severe acute or chronic medical or psychiatric condition or laboratory abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged 18 years and over diagnosed with stage IIIb/IV non-squamous NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Concordance in the detection of molecular abnormalities using Inivata liquid biopsy panel with detection using standard of care tissue biopsy analysis. | 12 months
  The primary endpoint is concordance in detecting molecular abnormalities using Inivata liquid biopsy panel compared with detection using tissue biopsy analysis.

SECONDARY OUTCOMES:
Sensitivity of Inivata liquid biopsy analysis relative to matched tissue analysis | 12 months
  Detection of sensitivity of molecular abnormalities using Inivata liquid biopsy panel relative to standard of care tissue biopsy analysis
Specificity of Inivata liquid biopsy analysis relative to matched tissue analysis | 12 months
  Detection of specificity of molecular abnormalities using Inivata liquid biopsy panel relative to standard of care tissue biopsy analysis
Description of the ctDNA profile of genomic alterations in patients where tumour tissue is limited versus that observed where tumour biopsy is achieved | 12 months
  Description of the ctDNA profile of genomic alterations in patients where tumour tissue is limited (Quantity Not Sufficient) versus that observed where tumour biopsy is achieved.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mercy Hospital Cancer Center/Clinical Research, Fort Smith, Arkansas
  - Mercy Cancer Center, Joplin, Missouri
  - Mercy Clinic, Springfield, Missouri
  - Mercy Clinic Oncology & Hematology, Oklahoma City, Oklahoma
  - Lehigh Valley Health Networks, Allentown, Pennsylvania
  - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: No